CLINICAL TRIAL: NCT03078400
Title: An Open-label Phase 1 Trial of the Safety and Efficacy of Daily Subcutaneous SPL-108 Injections When Used In Combination With Paclitaxel In Patients With Platinum-resistant, CD44+, Advanced Ovarian Epithelial Cancer
Brief Title: Safety and Efficacy Study of Daily SPL-108 Injections In Conjunction With Paclitaxel in Women With Ovarian Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Splash Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPL-006
Record Dates: First submitted 2017-03-04; First posted 2017-03-13 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Intervention Model Description: Arm I: N=6 to 12, Safety Phase, 3 + 3 design with 2 cohorts.
  * Cohort 1 SPL-108 150 mg daily + 80 mg/m2 PTX weekly on Days 1, 8, and 15 in 28 day cycles
  * Cohort 2 SPL-108 300 mg daily (150 mg q12 hours) + 80 mg/m2 PTX weekly on Days 1, 8, and 15 in 28 day cycles
  Arm II: N=up to 12, Exploratory Expansion Phase
  • Cohort 3: SPL-108 daily dose (to be determined in Arm I) + 80 mg/m2 PTX weekly on Days 1, 8, and 15 in 28 day cycles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety Phase (Experimental): Six to 12 subjects
  * Cohort 1 SPL-108 injection daily + 80 mg/m2 PTX weekly on Days 1, 8, and 15 in 28 day cycles
  * Cohort 2 SPL-108 BID injection + 80 mg/m2 PTX weekly on Days 1, 8, and 15 in 28 day cycles
  Interventions: Drug: SPL-108
- Exploratory Expansion Phase (Experimental): Up to 12 subjects
  • Cohort 3: SPL-108 daily dose (to be determined in Arm I) + 80 mg/m2 PTX weekly on Days 1, 8, and 15 in 28 day cycles.
  Interventions: Drug: SPL-108

INTERVENTIONS:
Drug: SPL-108 — Subcutaneous injection of 150 mg administered either one time or two times per day.

SUMMARY:
Up to 18 women with ovarian cancer will administer up to two injections of SPL-108 daily in combination with weekly doses of Paclitaxel. They will be monitored for safety and efficacy for up to 6 months, until disease progression or unacceptable toxicity.

DETAILED DESCRIPTION:
This is an open-label 2-arm trial. Eligible subjects will be screened and enrolled sequentially into 1 of 2 Arms:

Arm I: N=6 to 12 subjects, Safety Phase

* Cohort 1 SPL-108 x 1 injection daily + 80 mg/m2 PTX weekly on Days 1, 8, and 15 in 28 day cycles
* Cohort 2 SPL-108 BID + 80 mg/m2 PTX weekly on Days 1, 8, and 15 in 28 day cycles

For Arm I, at least 1 week will elapse between Dose 1 for each subject.

In Cohort 1, 3 subjects will be enrolled: if 1 dose-limiting toxicity (DLT) occurs, 3 subjects will be added at this dose level; if 0/3 or 1/6 DLTs occur, Cohort 2 will initiate enrolling subjects; if 2 or more DLTs occur at this dose level, subjects will not be enrolled in Cohort 2 and the trial will be terminated.

In Cohort 2, 3 subjects will be enrolled: if 1 DLT occurs, 3 subjects will be added at this dose level; if 0/3 or 1/6 DLTs occur, Arm II will initiate enrolling subjects at the SPL-108 BID dose; if 2 or more DLTs occur, Arm II will initiate enrolling subjects at the SPL-108 dose one time each day.

Arm II: N=up to 12, Exploratory Expansion Phase

• Cohort 3: SPL-108 daily dose (to be determined in Arm I) + 80 mg/m2 PTX weekly on Days 1, 8, and 15 in 28 day cycles.

A Safety Committee will meet at the end of each Arm I Cohort as well as periodically to review safety data and make recommendations for trial progression. The primary efficacy outcome, Response Evaluation Criteria in Solid Tumors Committee (RECIST 1.1) criteria, will be assessed on Day 15 of Cycles 2, 4, and 6.

ELIGIBILITY:
Inclusion Criteria:

1. Females ≥18 years of age
2. Platinum-resistant recurrent or metastatic epithelial ovarian carcinoma
3. Positivity on CD44 assay as defined by strong (+++) or moderate (++) staining in 20% or more of the tumor tissue/stroma as obtained by biopsy or paracentesis
4. Status post first-line therapy with definitive surgery (which provided tissue for pathologic diagnosis) and chemotherapy
5. Original diagnosis has been confirmed through a histopathologic review of the primary tumor slides by an expert pathologist at the Principal Investigator's institution
6. Disease has progressed or recurred during or less than 6 months after platinum-based chemotherapy at some point during the subject's course.
7. No more than 3 prior regimens of cytotoxic chemotherapy unless approved by the sponsor (Note: all platinum-containing regimens are not to be counted separately but are considered to be a single regimen for the purposes of this criterion)
8. Measurable disease by RECIST 1.1 criteria
9. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0, 1, or 2
10. Women with childbearing potential and partners must both use effective contraception during the study and for 3 months after the last dose
11. Life expectancy of at least 6 months
12. Able to understand and comply with the study procedures, understand the risks involved in the study, and provide written informed consent before the first study-specific procedure

Exclusion Criteria:

1. Treatment with cytotoxic chemotherapy for malignancies other than ovarian cancer within the past 5 years
2. Fewer than 28 days before Cycle 1 Day 1 since any prior chemotherapy (less than 42 days in the case of mitomycin or a nitrosourea)
3. Fewer than 28 days before Cycle 1 Day 1 since administration of hormonal or biological anti-neoplastic agents
4. Concomitant use of other cytotoxic or cytostatic drugs other than PTX
5. Abnormal clinical laboratory values within 14 days prior to initiation of dosing, as indicated by:

   * Hemoglobin level <9.0 gm/L
   * Platelet count <100,000/mm3
   * Granulocyte count <1500/mm3
   * Serum creatinine level ≥2.5 mg/dL (221 μmol/L)
   * Liver aminotransferase levels greater than 3 times the laboratory's upper limit of normal (greater than 5 times the laboratory's upper limit of normal if the liver is known to be involved with tumor)
6. Contraindication to the use of PTX
7. Pregnancy or breast-feeding at time of Screening and throughout the study.
8. Active, uncontrolled infection
9. Participation in another investigational drug trial concurrently or within 30 days of Cycle 1 Day 1, or a vaccine trial within 90 days of Cycle 1 Day 1
10. Significant acute or chronic medical or psychiatric illness that, in the judgment of the Investigator, could compromise subject safety, limit the subject's ability to complete the trial, and/or compromise the objectives of the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with advanced ovarian epithelial cancer
Enrollment: 14 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (Safety) | Until dose-limiting toxicity, disease progression or 6 months
  Includes adverse events, laboratory data, physical examination findings, vital signs, weight and ECOG Performance Status

SECONDARY OUTCOMES:
Response to Investigational Product | Until dose-limiting toxicity, disease progression or 6 months
  Objective response (OR) through imaging assessments
Response to Investigational Product | Until dose-limiting toxicity, disease progression or 6 months
  Objective response (OR) through changes in CA 125 levels
Response to Investigational Product | Until dose-limiting toxicity, disease progression or 6 months
  Objective response (OR) as assessed through changes in Quality of Life (FACT-O Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: June Girda, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Girda E, Hou J, Nelson D, Finlayson M, de Meritens AB, Chekmareiva M, Leiser A, Song M, Stephenson R, Chan N, Tergas AI, Vattakalam R, Wright JD, Yu H, Martincuks A, Kohut A, Palmer J, Rodriguez-Rodriguez L. Phase I trial of daily subcutaneous SPL-108 injections in combination with paclitaxel in patients with platinum resistant CD44+ advanced ovarian epithelial cancer. Int J Gynecol Cancer. 2022 Aug 1;32(8):1032-1038. doi: 10.1136/ijgc-2021-003316. PMID 35750354